CLINICAL TRIAL: NCT02753218
Title: LEO 32731 - A Phase I Drug-Drug Interaction Study With LEO 32731 and Midazolam in Healthy Male Subjects
Brief Title: A Phase I Study With LEO 32731 and Midazolam in Healthy Male Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to tolerability issues related to the dose titration, unexpected withdrawals were observed and it was unlikely for the trial to meet its objectives
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LP0058-1267
Record Dates: First submitted 2016-04-12; First posted 2016-04-27 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Midazolam and LEO 32731 (Experimental)
  Interventions: Drug: Midazolam; Drug: LEO 32731

INTERVENTIONS:
Drug: Midazolam
Drug: LEO 32731

SUMMARY:
The purpose of this study is to investigate the effects of multiple oral doses of LEO 32731 on the pharmacokinetics of a single oral dose of the cytochrome P450 3A substrate midazolam in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will, prior to any study-related activities, have given their written informed consent to participate in the study and to abide by the study restrictions.
* caucasian
* between 18 and 59 years of age, inclusive
* Subjects will have a body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive.
* Subjects must be of good health

Exclusion Criteria:

* Male subjects who are not willing, or whose partners are not willing, to use appropriate contraception (such as condom with spermicidal foam/gel/film/cream/suppository), or who are not willing to refrain from donating sperm from the time of the first dose until 3 months after the final dosing occasion.
* Male subjects whose partners are of child bearing potential must also agree to use an additional highly effective method of contraception
* Subjects who have received any prescribed systemic or topical medication within 14 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
* Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the first dose administration of midazolam.
* Subjects who have received any medications, including St John's Wort (or other dietary restriction), known to chronically alter drug absorption or elimination processes (change enzyme levels) within 30 days of the first dose administration of midazolam.
* Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity) or a marketed drug within the past 3 months prior to the first dosing occasion.
* Subjects who have donated any blood, plasma or platelets in 3 months prior to screening or who have made donations on more than 2 occasions within the 12 months preceding the first dose administration of midazolam.
* Subjects with a significant history of drug allergy as determined by the Investigator.
* Subjects who have any clinically significant allergic disease (excluding non-active hayfever) as determined by the Investigator.
* Subjects who have a supine blood pressure and supine pulse rate at screening higher than 140/90 mmHg and 100 beats per minute (bpm), respectively, or lower than 90/50 mmHg and 45 bpm, respectively.
* Subjects who consume more than 28 units of alcohol per week.
* Subjects who have a significant history of alcoholism or drug/chemical abuse as determined by the Investigator.
* Subjects with a positive urine drugs of abuse screen or alcohol breath test result at screening or first admission.
* Subjects who smoke or who have smoked in the 3 months prior to first dose administration.
* Subjects with, or with a history of, any clinically significant neurological, gastrointestinal (GI), renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological, dermatological or other major disorders as determined by the Investigator.
* Subjects who have had a clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator.
* Subjects who are known to have serum hepatitis, or who are carriers of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody, or who have a positive result to the test for human immunodeficiency virus (HIV) antibodies.
* Active tuberculosis or history of incompletely treated tuberculosis, based on medical history or medical report, or tuberculosis test at screening.
* Subjects who, in the opinion of their General Practitioner or the Investigator, should not participate in the study, including subjects suspected for whatever reason of not being able to comply with the requirements of the protocol.
* Subjects who have an abnormality in the 12-lead ECG that, in the opinion of the Investigator, increases the risk of participating in the study.

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of midazolam on Day 17 | 17 days
Peak Plasma Concentration (Cmax) of midazolam on Day 17 | 17 days

SECONDARY OUTCOMES:
AUC of midazolam on Day 1 | 1 day
Cmax of midazolam on Day 1 | 1 day
Incidence and severity of adverse events (AEs) defined as spontaneously reported AEs and clinically significant values reported as AEs | 54 days
  Assessments for: blood pressure, pulse, temperature, pulse oximetry, 12-lead electrocardiograms (ECGs), physical examinations, and laboratory evaluations

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Ltd., Springfield House, Hyde Street, Leeds, United Kingdom